CLINICAL TRIAL: NCT05482685
Title: The Health-Promoting Behavior and Related Factors Among Home Care Attendants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202206098RINB
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Health Promotion
Keywords: home care attendant; health-promoting behavior; health literacy; self-perceived health
MeSH Terms: conditions — Health Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Demographic variables: Include gender, age, BMI, education level, marital status, attended health promotion program or not, average monthly income, years of experience, average hours of work per week, chronic illness, smoking habit, drinking habit
  Interventions: Behavioral: Questionnaire
- health literacy: The number of points scored by completing the scale
  Interventions: Behavioral: Questionnaire
- self-perceived health: The number of points scored by completing the scale
  Interventions: Behavioral: Questionnaire
- health-promoting behavior: The number of points scored by completing the scale
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Conduct a 10-minute survey

SUMMARY:
Background: With the trend of aging population and increasing demand for long-term care, Taiwan's long-term care 2.0 policy places special emphasis on home care services to achieve the goal of local aging. This study focused on the health-promoting behaviors home care attendants and applied Pender's health promotion model theory to investigate the impact of home care attendants' self-perceived health and health literacy on health-promoting behaviors.

Objective: To investigate the current status of home care attendants' health-promoting behaviors and the correlation between self-perceived health and health literacy.

Methodology: A structured questionnaire was used to collect data from 150 eligible home care attendants in the northern region using self-perceived health, health literacy, and health-promoting behaviors scales. Multiple regression analysis was used to analyze the correlation between the independent variables and the dependent variables.

Expected contribution: The results of this study will help to understand the current status of health-promoting behaviors of home care attendants and the correlation with their self-perceived health and health literacy. It will also help to understand whether home care attendants have sufficient health literacy to maintain or improve their health status, and to understand the areas in which home care attendants' health-promoting behaviors are still inadequate, so as to suggest effective methods or strategies to improve health-promoting behaviors in the future.

ELIGIBILITY:
Inclusion Criteria:

1. have license or have received training and a certificate of completion.
2. have been working in home care for at least three months
3. agree to participate in the study.

Exclusion Criteria:

1. under 20 years of age.
2. non-national.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: home care attendants
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Survey questionnaire | 10 minutes
  Understand the current status of health-promoting behaviors of home care attendants and the correlation with their self-perceived health and health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Ku Shan-Ting, bachelor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No